CLINICAL TRIAL: NCT00068224
Title: Clinical and Molecular Investigations Into Ciliopathies
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030264; 03-HG-0264
Record Dates: First submitted 2003-09-10; First posted 2003-09-10 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Ciliopathy
Keywords: Caroli's Syndrome; Congenital Hepatic Fibrosis; Ductal Plate Malformation; Polycystic Kidney; Autosomal Recessive Polycystic Kidney Disease; ARPKD; Kidney; Liver
MeSH Terms: conditions — Ciliopathies; Caroli Disease; Hepatic Fibrosis, Congenital; Polycystic Kidney Diseases; Polycystic Kidney, Autosomal Recessive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ciliopathy: Children and adults who carry a clinical diagnosis of a known ciliopathy and those patients who have typical features suggestive of a cliopathy but not fulfilling the diagnostic criteria.

SUMMARY:
This study will evaluate patients ciliopathies. People with ciliopathies develop fibrocystic disease of the kidneys and liver, retinal degeneration, obesity, structural and functional defects of the central nervous system and the eyes, abnormal bone growth, abnormal sidedness of internal organs and polydactyly. The goal of the study is to better understand the medical complications of these disorders and identify characteristics that can help in the design of new treatments.

DETAILED DESCRIPTION:
Human diseases caused by defects of the primary cilium (ciliopathies) are a group of distinct disorders with overlapping features. Clinical features of ciliopathies include fibrocystic disease of the kidneys and liver, retinal degeneration, obesity, structural and functional defects of the central nervous system and the eyes, abnormal bone growth, abnormal sidedness of internal organs and polydactyly. Human ciliopathies characterized by variable combinations of these features include autosomal recessive (ARPKD) and dominant (ADPKD) polycystic kidney diseases, nephronophthisis (NPHP), Joubert syndrome and related disorders (JSRD), Bardet-Biedl (BBS), Meckel-Gruber (MKS), Oral-Facial-Digital-type 1 (OFD1), and Alstrom syndromes (AS) and skeletal disorders such as Jeune syndrome (JS) and cleidocranial dysplasia. ARPKD, the most common pediatric ciliopathy, is characterized by cystic degeneration of the kidneys and congenital hepatic fibrosis of the liver. JSRD are a heterogenous group of syndromes characterized by a distinctive cerebellar and brainstem malformation (molar tooth sign), intellectual disability, abnormal eye movements, and abnormal respiratory pattern in infancy. Other common features seen in subsets of JSRD patients include, fibrocystic renal disease, congenital hepatic fibrosis, retinal degeneration, retinal colobomas, occipital encephalocele, and polydactyly. AS and BBS are ciliopathies characterized by obesity and retinal degeneration and hepatorenal disease in most cases. BBS patients also exhibit postaxial polydactyly, cognitive impairment, male hypogonadotrophic hypogonadism and female genitourinary malformations. Additional features in AS include metabolic syndrome associated with insulin resistance and hyperlipidemia, cardiomyopathy and sensorineural deafness. OFD-I is characterized by polycystic kidney disease and oral, digital and brain anomalies including cerebellar hypoplasia with or without Dandy-Walker malformation. JS is a skeletal ciliopathy characterized by small thorax, short-limbed short stature, fibrocystic renal disease and retinal degeneration. The frequency and characteristics and natural history of specific organ/system disease in ciliopathies are either unknown or poorly defined, mostly because of the limited data available from retrospective reports of small numbers of patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Children and adults who carry a clinical diagnosis of a known ciliopathy such as ARPKD, CHF, JSRD, BBS, OFD1, AS and those patients who have typical features suggestive of a ciliopathy but not fulfilling the diagnostic criteria for any

of the known disorders (unknown types of PKD and/or CHF, retinal degeneration, variants of molar tooth sign such as Dandy-Walker variants). This might rarely include adults who are unable to give informed consent.

Among patients who have received a kidney or liver allograft, those with stable graft function and without severe transplantrelated

complications are eligible for enrollment.

EXCLUSION CRITERIA:

Infants under 6 months of age

Medically fragile patients who require frequent hospitalizations due to complications of end-stage renal disease (uncontrolled hypertension, severe electrolyte imbalances), hepatic disease (current variceal bleeding, overt encephalopathy, intractable recurrent cholangitis), severe cardiomyopathy as seen in some AS patients, or severe respiratory abnormalities as seen in some JSRD patients with severe brain stem involvement.

Ages: 5 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults who carry a clinical diagnosis of a known ciliopathy such as ARPKD, CHF, JSRD, BBS, OFD1, AS and those patients who have typical features suggestive of a ciliopathy but not fulfilling the diagnostic criteria for any of the known disorders (unknown types of PKD and/or CHF, retinal degeneration, variants of molar tooth sign such as Dandy-Walker variants).
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2003-03-16 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Ciliopathy | ongoing
  The general objective of this study is to assess the clinical characteristics of ciliopathies.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Gunay-Aygun, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gunay-Aygun M, Font-Montgomery E, Lukose L, Tuchman M, Graf J, Bryant JC, Kleta R, Garcia A, Edwards H, Piwnica-Worms K, Adams D, Bernardini I, Fischer RE, Krasnewich D, Oden N, Ling A, Quezado Z, Zak C, Daryanani KT, Turkbey B, Choyke P, Guay-Woodford LM, Gahl WA. Correlation of kidney function, volume and imaging findings, and PKHD1 mutations in 73 patients with autosomal recessive polycystic kidney disease. Clin J Am Soc Nephrol. 2010 Jun;5(6):972-84. doi: 10.2215/CJN.07141009. Epub 2010 Apr 22. PMID 20413436
- [Background] Gunay-Aygun M. Liver and kidney disease in ciliopathies. Am J Med Genet C Semin Med Genet. 2009 Nov 15;151C(4):296-306. doi: 10.1002/ajmg.c.30225. PMID 19876928
- [Background] Gunay-Aygun M, Font-Montgomery E, Lukose L, Tuchman Gerstein M, Piwnica-Worms K, Choyke P, Daryanani KT, Turkbey B, Fischer R, Bernardini I, Sincan M, Zhao X, Sandler NG, Roque A, Douek DC, Graf J, Huizing M, Bryant JC, Mohan P, Gahl WA, Heller T. Characteristics of congenital hepatic fibrosis in a large cohort of patients with autosomal recessive polycystic kidney disease. Gastroenterology. 2013 Jan;144(1):112-121.e2. doi: 10.1053/j.gastro.2012.09.056. Epub 2012 Oct 3. PMID 23041322
- [Derived] Brooks BP, Zein WM, Thompson AH, Mokhtarzadeh M, Doherty DA, Parisi M, Glass IA, Malicdan MC, Vilboux T, Vemulapalli M, Mullikin JC, Gahl WA, Gunay-Aygun M. Joubert Syndrome: Ophthalmological Findings in Correlation with Genotype and Hepatorenal Disease in 99 Patients Prospectively Evaluated at a Single Center. Ophthalmology. 2018 Dec;125(12):1937-1952. doi: 10.1016/j.ophtha.2018.05.026. Epub 2018 Jul 25. PMID 30055837
- [Derived] Han JC, Reyes-Capo DP, Liu CY, Reynolds JC, Turkbey E, Turkbey IB, Bryant J, Marshall JD, Naggert JK, Gahl WA, Yanovski JA, Gunay-Aygun M. Comprehensive Endocrine-Metabolic Evaluation of Patients With Alstrom Syndrome Compared With BMI-Matched Controls. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2707-2719. doi: 10.1210/jc.2018-00496. PMID 29718281
- [Derived] Boerwinkle C, Marshall JD, Bryant J, Gahl WA, Olivier KN, Gunay-Aygun M. Respiratory manifestations in 38 patients with Alstrom syndrome. Pediatr Pulmonol. 2017 Apr;52(4):487-493. doi: 10.1002/ppul.23607. Epub 2016 Dec 28. PMID 28029746
- [Derived] Vilboux T, Malicdan MC, Chang YM, Guo J, Zerfas PM, Stephen J, Cullinane AR, Bryant J, Fischer R, Brooks BP, Zein WM, Wiggs EA, Zalewski CK, Poretti A, Bryan MM, Vemulapalli M, Mullikin JC, Kirby M, Anderson SM; NISC Comparative Sequencing Program; Huizing M, Toro C, Gahl WA, Gunay-Aygun M. Cystic cerebellar dysplasia and biallelic LAMA1 mutations: a lamininopathy associated with tics, obsessive compulsive traits and myopia due to cell adhesion and migration defects. J Med Genet. 2016 May;53(5):318-29. doi: 10.1136/jmedgenet-2015-103416. Epub 2016 Jan 13. PMID 27095636
- [Derived] Malicdan MC, Vilboux T, Stephen J, Maglic D, Mian L, Konzman D, Guo J, Yildirimli D, Bryant J, Fischer R, Zein WM, Snow J, Vemulapalli M, Mullikin JC, Toro C, Solomon BD, Niederhuber JE; NISC Comparative Sequencing Program; Gahl WA, Gunay-Aygun M. Mutations in human homologue of chicken talpid3 gene (KIAA0586) cause a hybrid ciliopathy with overlapping features of Jeune and Joubert syndromes. J Med Genet. 2015 Dec;52(12):830-9. doi: 10.1136/jmedgenet-2015-103316. Epub 2015 Sep 18. PMID 26386044
- [Derived] Banks N, Bryant J, Fischer R, Huizing M, Gahl WA, Gunay-Aygun M. Pregnancy in autosomal recessive polycystic kidney disease. Arch Gynecol Obstet. 2015 Mar;291(3):705-8. doi: 10.1007/s00404-014-3445-8. Epub 2014 Sep 12. PMID 25214022
- [Derived] O'Brien K, Font-Montgomery E, Lukose L, Bryant J, Piwnica-Worms K, Edwards H, Riney L, Garcia A, Daryanani K, Choyke P, Mohan P, Heller T, Gahl WA, Gunay-Aygun M. Congenital hepatic fibrosis and portal hypertension in autosomal dominant polycystic kidney disease. J Pediatr Gastroenterol Nutr. 2012 Jan;54(1):83-9. doi: 10.1097/MPG.0b013e318228330c. PMID 21694639
- [Derived] Gunay-Aygun M, Parisi MA, Doherty D, Tuchman M, Tsilou E, Kleiner DE, Huizing M, Turkbey B, Choyke P, Guay-Woodford L, Heller T, Szymanska K, Johnson CA, Glass I, Gahl WA. MKS3-related ciliopathy with features of autosomal recessive polycystic kidney disease, nephronophthisis, and Joubert Syndrome. J Pediatr. 2009 Sep;155(3):386-92.e1. doi: 10.1016/j.jpeds.2009.03.045. Epub 2009 Jun 21. PMID 19540516
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-HG-0264.html